CLINICAL TRIAL: NCT02417532
Title: Safety and Feasibility Evaluation of Robot Assisted Physiotherapy Exercises With REX
Acronym: RAPPER II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rex Bionics Plc (Industry)
Collaborators: Generic Devices Consulting, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RXPR-0001
Record Dates: First submitted 2015-04-11; First posted 2015-04-15 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rehabilitation using REX (Experimental): Exercises using Rex mobility assist device
  Interventions: Device: Rehabilitation using REX

INTERVENTIONS:
Device: Rehabilitation using REX — Exercises of wheelchair dependent subjects using REX

SUMMARY:
Prospective, Open label, single arm, non-randomized, non-comparative registry study of Robot-Assisted Physiotherapy Exercises with the REX Robot powered exercise system in patients with Spinal cord or other injury preventing unsupported patient ambulation.

DETAILED DESCRIPTION:
The objective of this feasibility study is to evaluate the overall device safety when used in Spinal Cord Injury Hospitals or Rehabilitation Centers under the supervision of a physician and/or qualified rehabilitation specialists.

ELIGIBILITY:
Inclusion Criteria

* Wheelchair user
* Spinal Injury Levels of C4 down to L5
* Has no outstanding skin integrity issues that could be effected by the REX device
* Should be between approximately 1.42m and 1.93m in height. More specifically, REX is able to accommodate the following limb lengths:
* Upper leg length : 380 - 470 mm
* Lower leg length : 366 - 470 mm
* Heel position (Ankle to hind foot) : 40 - 92 mm
* Floor to ankle height (To be measured while wearing the shoe to be used for mobilising in REX) : 96 - 116 mm
* Has a skeletal hip width of 380 mm or less (limit imposed by REX)
* Is between 40 kg and 100 kg weight (limits imposed by REX)
* Has the manual dexterity to work a joystick
* Sufficient passive range of motion in the Hip, Knee and Ankle of at least
* Hip 90 degrees flexion 15 degrees hip extension 20 degrees abduction 16 degrees adduction
* Knee 0 degrees extension 93 degrees flexion
* Ankle 20 degrees dorsiflexion (with weight bearing and 10 degrees knee flexion) 22 degrees dorsiflexion (with 93 degrees knee flexion) 10 degrees plantar flexion 9 degrees inversion 9 degrees eversion
* Thigh lateral diameter of < 135 mm (230 mm above the knee joint line)
* Calf lateral diameter of < 100 mm (90 mm below the knee joint line)
* Manual dexterity to work a joystick with or without a T-Bar and use emergency stop button
* No contraindications to standing or mobilising
* Patients must choose to participate, and must have signed the informed consent document

Exclusion Criteria:

* Patients who do not meet inclusion criteria or physician discretion.
* Patients with history of impaired cardiac function who have been referred to and reviewed by a medical professional. With a decision made that they should not continue in the trial due to their impaired cardiac function.
* Patients contraindicated to walk or stand
* Patients with spinal injury outside Inclusion criteria
* Withdrawal or refusal to sign informed consent
* Any other contraindication based on physician discretion
* Known allergy (skin contact) to materials used in Rex

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Birch, FRCS, Principal Investigator — The Chris Moody Centre
Locations (6):
- Austin Health, Heidelberg, Victoria, Australia
- New Zealand (2):
  - Rehabilitation Innovation Centre at AUT University, Auckland
  - Canterbury District Health Board, Burwood Hospital, Christchurch
- United Kingdom (3):
  - East Kent Hospitals University Foundation Trust, Canterbury, Kent
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore, Middlesex
  - Physiofunction, Moulton, Northamptonshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birch N, Graham J, Priestley T, Heywood C, Sakel M, Gall A, Nunn A, Signal N. Results of the first interim analysis of the RAPPER II trial in patients with spinal cord injury: ambulation and functional exercise programs in the REX powered walking aid. J Neuroeng Rehabil. 2017 Jun 19;14(1):60. doi: 10.1186/s12984-017-0274-6. PMID 28629390

RESULTS

PARTICIPANT FLOW:
Groups:
- Rex Rehabilitation Patients: Tetraplegic and paraplegic patients able to use REX.
Period: Overall Study
Arm/Group | Rex Rehabilitation Patients
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants] — Age - from date of birth record
  Participants
    <=18 years | 1
    Between 18 and 65 years | 54
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 39.8 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 37
Region of Enrollment [Number; unit: participants]
  New Zealand | 3
  United Kingdom | 9
  Australia | 44

OUTCOME MEASURES:

1. Primary Outcome: Ability to Transfer
Description: Completion of transfer with supervision or 1 assistant from wheelchair or bed into REX
Time Frame: 1 day
Population: All subjects meeting inclusion criteria. Physically able to properly fit in REX.
Measure: Number; unit: participants
Groups:
- Rehabilitation Using REX: Tetraplegic and paraplegic patients
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 56
participants | 32

2. Primary Outcome: Adverse Events
Description: absence of unexpected serious adverse events
Time Frame: 1 day
Population: All patients transferring into Rex.
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 56
Participants | 56

3. Primary Outcome: Transfer Time
Description: Time it took for participant to transfer into the Rex with or without supervision.
Time Frame: 1 day
Population: All patients transferring into Rex
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 56
seconds | 352.2 (75)

4. Secondary Outcome: Participant Satisfaction Questionnaire
Description: overall user satisfaction with the device
Time Frame: 1 Day
Population: Patients who were able to transfer into REX and who could control the joystick. One patient was unable to walk and control Rex so did not complete the questionaire.
Measure: Number; unit: percentage of patients
Groups:
- Rehabilitation Using REX: Tetraplegic and paraplegic patients who could control REX
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 55
percentage of patients
  Easy to Transfer % positive | 57
  Confidence % positive | 91
  Safety % positive | 88
  Stability % positive | 89
  Ease of control % positive | 84
  Comfort % positive | 84
  Wellbeing following use % positive | 82
  Benefits to using regularly % positive | 91
  The size of REX did not bother me | 64
  The sound of REX did not bother me % positive | 73
  The speed of REX was suitable for me % positive | 61

5. Secondary Outcome: Timed up and go Test- Ability to Stand From Chair
Description: The number of seconds required to walk 3 m and turn around and walk back to the chair. (Functional test)
Time Frame: 1 Day
Population: Subjects who were able to control the joystick. One patient was unable to control the joystick and was excluded.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rehabilitation Using REX
Number analyzed (Participants) | 55
seconds | 316.41 (91.52)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Rehabilitation Using REX: All patients who were able to transfer into a Rex with or without assistance.
Arm/Group | Rehabilitation Using REX
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

LIMITATIONS AND CAVEATS:
Patients enrolled under at different times in the recruitment process had differing lengths of follow-up as reflected in the final study report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No